CLINICAL TRIAL: NCT00808418
Title: A Phase 1 Study of Weekly Elesclomol Sodium Plus Docetaxel and Concomitant Prednisone in Subjects With Metastatic Castration Refractory Prostate Cancer (m-CRPC)
Brief Title: A Study to Determine the Maximum Tolerated Dose of Elesclomol Sodium Given With a Fixed Dose of Docetaxel and Prednisone in Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4783-12
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Prostate Cancer
Keywords: prostate; cancer; metastatic; castration; refractory; elesclomol; sodium; docetaxel; prednisone
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort (Experimental)
  Interventions: Drug: Elesclomol Sodium; Drug: Docetaxel

INTERVENTIONS:
Drug: Elesclomol Sodium — Chemotherapy agent
Drug: Docetaxel — Chemotherapy agent

SUMMARY:
This aim of this study is to determine the safety and tolerability of elesclomol sodium at escalating doses (ultimately identifying the maximum tolerated dose) when combined with a fixed dose of docetaxel and concomitant prednisone. This study will also characterize the pharmacokinetics of elesclomol and docetaxel.

DETAILED DESCRIPTION:
This aim of this study is to determine the safety and tolerability of elesclomol sodium at escalating doses (ultimately identifying the maximum tolerated dose) when combined with a fixed dose of docetaxel and concomitant prednisone. This study will also characterize the pharmacokinetics of elesclomol and docetaxel.

ELIGIBILITY:
Inclusion Criteria

* Confirmed metastatic prostate cancer
* No more than one prior chemotherapy on which the disease progressed
* ECOG performance status of less than or equal to 2
* Adequate bone marrow, renal and hepatic functions as defined in the protocol
* Neuropathy less than or equal to 2
* Reliable venous access for frequent study drug infusions

Exclusion Criteria

* Significant cardiovascular disease
* Known active brain metastases
* Subjects that have received treatment for other malignancies with in the past 5 years
* Other clinically significant uncontrolled conditions

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To characterize the safety and tolerability of escalating doses of elesclomol sodium in combination with a fixed dose of docetaxel and concomitant prednisone administered weekly to m-CRPC subjects | Jan 2011
To determine the MTD of elesclomol sodium when administered with 30 mg/m2 weekly docetaxel | Jan 2011
To characterize the pharmacokinetics of elesclomol sodium and docetaxel in this population | Jan 2011

SECONDARY OUTCOMES:
To evaluate anti-tumor activity at the MTD in castration refractory prostate cancer | Jan 2011
Evaluate OS | Jan 2011
To characterize the pharmacokinetics of elesclomol metabolites | Jan 2011

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Pacific Coast Hematology/Oncology Medical Group, Fountain Valley, California
  - Mayo Clinic, Rochester, Maryland
  - Mid Dakota Clinic, Bismarck, North Dakota
  - University of Texas Health Science Center, Cancer Therapy & Research Center, Institute for Drug Development, San Antonio, Texas
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin